CLINICAL TRIAL: NCT04388735
Title: Quality of Life and Psychological Distress in Patients With Multiple Myeloma and Their Caregivers
Brief Title: Multiple Myeloma (MM) Quality of Life (QOL) Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Kully Family Foundation (Unknown)
Responsible Party: Principal Investigator, Elizabeth O'Donnell, Principal Investigator, Massachusetts General Hospital
Other Study IDs: 19-816
Record Dates: First submitted 2020-05-12; First posted 2020-05-14 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Multiple Myeloma; Quality of Life; Symptom, Behavioral
Keywords: Multiple Myeloma; Quality of Life; Symptom, Behavioral
MeSH Terms: conditions — Multiple Myeloma; Behavioral Symptoms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Newly Diagnosed MM 1st Line and Caregivers: This research study's procedures include screening for eligibility, participant designation of a caregiver and a series of questionnaires.
  * Patients will be asked to identify a caregiver (e.g. a relative or friend) upon whom they rely for help and has an in-person contact with the patient at least 2x per week.
  * Both patients with or without identified caregivers will complete a one time series of questionnaires.
    * The questionnaires are completed one time only and measure quality of life, mood, coping strategies, and prognostic understanding and can be completed in the hospital, clinic, over the email, or telephone with assistance provided as needed.Questionnaires take approximately 20 minutes to complete.
  Interventions: Behavioral: Questionnaire
- MM receiving 1-3 prior lines of therapy and Caregivers: This research study's procedures include screening for eligibility, participant designation of a caregiver and a series of questionnaires.
  * Patients will be asked to identify a caregiver (e.g. a relative or friend) upon whom they rely for help and has an in-person contact with the patient at least 2x per week.
  * Both patients with or without identified caregivers will complete a one time series of questionnaires.
    * The questionnaires are completed one time only and measure quality of life, mood, coping strategies, and prognostic understanding and can be completed in the hospital, clinic, over the email, or telephone with assistance provided as needed.Questionnaires take approximately 20 minutes to complete
  Interventions: Behavioral: Questionnaire
- MM patients receiving ≥ 4 lines of therapy and Cargivers: This research study's procedures include screening for eligibility, participant designation of a caregiver and a series of questionnaires.
  * Patients will be asked to identify a caregiver (e.g. a relative or friend) upon whom they rely for help and has an in-person contact with the patient at least 2x per week.
  * Both patients with or without identified caregivers will complete a one time series of questionnaires.
    * The questionnaires are completed one time only and measure quality of life, mood, coping strategies, and prognostic understanding and can be completed in the hospital, clinic, over the email, or telephone with assistance provided as needed.Questionnaires take approximately 20 minutes to complete
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Series of questions covering quality of life, physical and psychological symptom burden, mood, and illness and prognostic understanding administered in person or remotely.

SUMMARY:
The main purpose of this study is to examine differences in quality of life and psychological distress for both Multiple Myeloma patients receiving treatment and their caregivers and to assess patient and caregiver prognostic understanding (understanding of the likely course of a disease over time) of Multiple Myeloma to guide development of more personalized treatment plans.

This study looks to further understand quality of life changes throughout multiple myeloma therapy for both patients and caregivers to help determine ways to improve patient and caregiver understanding of illness and in turn, tailor customized treatment that best aligns with patient preferences.

The study will use a series of questionnaires to measure quality of life, mood, coping strategies, and prognostic understanding.

DETAILED DESCRIPTION:
This research study's procedures include screening for eligibility, participant designation of a caregiver and a series of questionnaires.

- It is expected that about 180 people undergoing treatment for multiple myeloma and up to 180 of their caregivers will take part in this research study.

-- The questionnaires are completed one time only and measure quality of life, mood, coping strategies, and prognostic understanding and can be completed in the hospital, clinic, over the email, or telephone with assistance provided as needed.Questionnaires take approximately 20 minutes to complete.

ELIGIBILITY:
Inclusion Criteria:

Patient Eligibility criteria:

* Adult patients (greater than 18 years) receiving active therapy for MM.

  * For patients with newly diagnosed MM, patients are eligible while undergoing induction therapy prior to received autologous stem cell transplant but not after.
* Ability to read questions in English or willing to complete questionnaires with the assistance of an interpreter.

Caregiver Eligibility criteria:

* Adult (greater than 18 years) relative or a friend of a patient who agrees to participate in the study whom the patient identified as living with them or having in-person contact with him or her at least twice per week.
* Ability to read and respond to questions in English or to complete questionnaires with minimal assistance of an interpreter

Exclusion Criteria:

* Patient Exclusion criteria:

  * Patients receiving maintenance therapy only.
  * Significant psychiatric or other co-morbid disease, which the treating clinician believes prohibits informed consent or participation in the study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients receiving therapy for Multiple Myeloma and their identified/designated caregivers.
Sampling Method: Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2021-11-15 (Estimated); Study Completion 2022-05-16 (Estimated)

PRIMARY OUTCOMES:
Quality of life (QOL) Patient Description | Up to 1 year
  Describe patient QOL scores by lines of therapy. Functional Assessment of Cancer Therapy-Multiple Myeloma(FACT-MM) will be used to assess QOL, which has been validated for use in multiple care settings.[10]. The FACT-MM consists of four subscales assessing well-being across four domains (physical, functional, emotional, and social). These self-reported measures possess strong psychometric properties and have been validated for patients with cancer [Appendix E].
Quality of life (QOL) Caregiver Description | Up to 1 year
  Describe cargiver QOL scores by associated patient line of therapy

SECONDARY OUTCOMES:
QOL-Functional Assessment | Up to 1 year
  Describe and compare patient QOL Functional Assessment of Cancer Therapy-Multiple Myeloma (FACT-MM) scores by line of therapy. The FACT-MM consists of four subscales assessing well-being across four domains (physical, functional, emotional, and social). These self-reported measures possess strong psychometric properties and have been validated for patients with cancer
Patient Burden Assessment-ESAS | Up to 1 year
  Describe and compare patient symptoms (ESAS) scores by line of therapy. The Edmonton Symptom Assessment System (ESAS) will be used to ascertain the symptom burden experienced by patients. This previously validated survey assesses nine symptoms frequently reported by patients with cancer: pain, tiredness, nausea, depression, anxiety, drowsiness, appetite, well-being, and shortness of breath [
Patient Fatigue Symptoms | Up to 1 year
  Describe and compare patient fatigue symptoms (FACIT-Fatigue) by line of therapy.
  The Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-Fatigue), a 13-item FACIT subscale specific to fatigue that measures an individual's level of fatigue during their usual daily activities over the past week.[13, 14] The level of fatigue is measured on a 4-point Likert scale .
Patient anxiety symptoms | Up to 1 year
  Describe and compare patient anxiety and depression symptoms Hospital Anxiety and Depression Scale (HADS) to assess symptoms of depression and anxiety in all study participants. The HADS is a 14-item questionnaire that contains two 7-item subscales assessing depression and anxiety symptoms during the past week.. Scores on each subscale range from 0 to 21, with a cutoff of 8 or greater denoting clinically significant anxiety or depression
Patient Depression symptoms | Up to 1 year
  Describe and compare patient anxiety and depression symptoms Hospital Anxiety and Depression Scale Hospital Anxiety and Depression Scale (HADS) to assess symptoms of depression and anxiety in all study participants. The HADS is a 14-item questionnaire that contains two 7-item subscales assessing depression and anxiety symptoms during the past week.. Scores on each subscale range from 0 to 21, with a cutoff of 8 or greater denoting clinically significant anxiety or depression
Patient Post-traumatic stress symptoms | Up to 1 year
  Describe and compare post-traumatic stress symptoms (PCL-C) by line of therapy The Post-Traumatic Stress Disorder Checklist (PCL) to assess symptoms of post-traumatic stress in patients and caregivers. The PCL is a 17 item self-reported measure that evaluates symptoms of post traumatic stress disorder according to the criteria of the Diagnostic and Statistical Manual of Mental Disorders-IV
Patient coping | Up to 1 year
  Describe and compare patient coping (Brief Cope) by line of therapy. The Brief Cope, a 28-item questionnaire that assess 14 methods of coping (e.g., self-distraction, humor, denial) using a 4-point Likert scale
Caregiver Quality of Life (QOL) | Up to 1 year
  Describe and compare caregiver burden and QOL (CARGOQOL) scores by line of therapy. CareGiver Oncology QOL questionnaire (CARGOQOL) will be used to measure caregiver QOL. The CarGOQOL is a 29-item well-validated instrument to measure QOL in multiple domains.
Caregiver Burden | Up to 1 year
  Describe and compare caregiver burden and QOL (CARGOQOL) scores by line of therapy. CareGiver Oncology QOL questionnaire (CARGOQOL) will be used to measure caregiver QOL. The CarGOQOL is a 29-item well-validated instrument to measure QOL in multiple domains.
Caregiver anxiety | Up to 1 year
  Describe and compare caregiver anxiety and depression symptoms (caregiver HADS) by line of therapy. The Hospital Anxiety and Depression Scale will be used to (HADS) to assess symptoms of depression and anxiety in all study participants (patients and family caregivers). The HADS is a 14-item questionnaire that contains two 7-item subscales assessing depression and anxiety symptoms during the past week. Scores on each subscale range from 0 to 21, with a cutoff of 8 or greater denoting clinically significant anxiety or depression
Caregiver Depression | Up to 1 year
  Describe and compare caregiver anxiety and depression symptoms (caregiver HADS) by line of therapy. The Hospital Anxiety and Depression Scale will be used to (HADS) to assess symptoms of depression and anxiety in all study participants (patients and family caregivers). The HADS is a 14-item questionnaire that contains two 7-item subscales assessing depression and anxiety symptoms during the past week. . Scores on each subscale range from 0 to 21, with a cutoff of 8 or greater denoting clinically significant anxiety or depression
Caregiver Coping | Up to 1 Year
  Describe and compare caregiver coping (Brief Cope) Brief Cope, a 28-item questionnaire that assess 14 methods of coping (e.g., self-distraction, humor, denial) using a 4-point Likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth K O'Donnell, MD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation